CLINICAL TRIAL: NCT00723554
Title: A Phase IIIb, Multicenter, Open-label Study of Patients With Pulmonary Arterial Hypertension Treated With Iloprost(Inhalation)Evaluating Safety and Inhalation Times When Converting From Power Disc-6 (PD-6) to Power Disc-15 (PD-15) With the I-neb® AAD®
Brief Title: Iloprost Power Disc-15 in Pulmonary Arterial Hypertension
Acronym: INHALE-15
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor's decision
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-063A402
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; inhaled therapy; power disc-15
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iloprost (Experimental): The study enrolled patients who were already using iloprost with PD-6 without any safety or tolerability concerns, thereby facilitating a direct comparison of the PD-15 to the PD-6.
  The single-arm design allowed each patient to serve as his/her own control
  Interventions: Drug: Iloprost PD-6; Drug: Iloprost PD-15

INTERVENTIONS:
Drug: Iloprost PD-6 — Period 1 (PD-6): study period defined as the 14 days prior to the first dose of study iloprost inhalation with PD-15. Commercial iloprost inhalation solution delivered using the Power Disc-6 with the I-neb® Adaptive Aerosol Delivery (AAD®) system administered 6 to 9 times per day
  Other Names: Ventavis
Drug: Iloprost PD-15 — Period 2 (PD-15): study period between the administration of the first dose with PD-15 on Day 1 until Day 28 inclusive.
  Period 3 (PD-15): study period from Day 29 until discontinuation of the PD-15. Commercial iloprost inhalation solution delivered using the Power Disc-15 with the I-neb® Adaptive Aerosol Delivery (AAD®) system administered 6 to 9 times per day
  Other Names: Ventavis

SUMMARY:
A Phase IIIb, Multicenter, Open-Label Study of Patients With Pulmonary Arterial Hypertension Treated With Iloprost(Inhalation)Evaluating Safety and Inhalation Times When Converting From Power Disc-6 to Power Disc-15 With the I-neb® Adaptive Aerosol Delivery® System (I-neb® AAD®)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-mandated procedure.
* Male or female patients aged 18-85 years.
* Patients with symptomatic pulmonary arterial hypertension in New York Heart Association (NYHA) functional class III or IV at the time of initiation of iloprost inhalation (Ventavis®) therapy using the Power Disc-6 (PD-6).
* Patients with the following types of pulmonary arterial hypertension (PAH) belonging to World Health Organization (WHO) Group I:

  * 1.1: Idiopathic (IPAH)
  * 1.2: Familial (FPAH)
  * 1.3: Associated with (APAH)

    * 1.3.1: Collagen vascular disease
    * 1.3.2: Congenital systemic-to-pulmonary shunts at least 2 years post surgical repair
    * 1.3.4: Human immunodeficiency virus (HIV) infection
    * 1.3.5: Drugs and toxins
* PAH confirmed by the most recent right heart catheterization showing:

  * Mean pulmonary arterial pressure (mPAP)≥ 25 mmHg at rest
  * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg. If both PCWP and LVEDP are available then the LVEDP value is retained for inclusion.
  * Pulmonary vascular resistance (PVR) > 240 dyn-sec/cm^5
* Compliant with a treatment regimen of commercial iloprost inhalation (Ventavis® 5 μg) using the I-neb® AAD® equipped with the PD-6 for at least 4 weeks prior to screening.
* Pulmonary function tests (PFTs) including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), and total lung capacity (TLC), performed within 6 months of screening.
* If taking other medications for PAH, these must have been stable for 60 days prior to baseline.
* If taking corticosteroids, these must have been stable for 60 days prior to baseline.
* Women of childbearing potential with a negative urine pre-treatment pregnancy test at baseline and who:

  * consistently and correctly use (from screening and up to 28 days after discontinuation of study drug) a reliable method of contraception with a Pearl index of < 1%,
  * are sexually abstinent, or
  * have a vasectomized partner.

A woman is considered to have childbearing potential unless she meets at least one of the following criteria:

* Previous bilateral salpingo-oophorectomy or hysterectomy
* Premature ovarian failure confirmed by a specialist gynecologist
* XY genotype, Turner syndrome, uterine agenesis
* Is aged > 50 years and not treated with any kind of hormone replacement therapy (HRT) for at least 2 years prior to screening, with amenorrhea for at least 24 consecutive months

Exclusion Criteria:

* PAH belonging to WHO group II-V.
* PAH belonging to WHO group I other than that listed in the inclusion criteria, i.e., PAH associated with:

  * 1.3.3: Portal hypertension
  * 1.3.6: Other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, splenectomy)
  * 1.4: Associated with significant venous or capillary involvement:

    * 1.4.1: Pulmonary veno-occlusive disease (PVOD)
    * 1.4.2: Pulmonary capillary hemangiomatosis (PCH).
* Receipt of any prostacyclin or prostacyclin analog other than iloprost within 12 weeks before screening.
* Anticipation of the need for intravenous prostacyclin use within 28 days of starting the Power Disc-15 (PD-15).
* HIV-seropositive with any of the following:

  * Concomitant active opportunistic infections within 6 months prior to screening
  * Detectable viral load within 6 months of screening
  * CD4+ T-cell count < 200 mm^3 within 3 months of screening
  * Changes in antiretroviral regimen within 3 months of screening
  * Anticipated changes in antiretroviral regimen during study periods 1 or 2
  * Using inhaled pentamidine
* Systemic hypotension with systolic blood pressure < 95 mmHg.
* Uncontrolled systemic hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg on repeated measurement).
* History of left-sided heart disease, including any of the following:

  * hemodynamically significant aortic or mitral valve disease
  * restrictive or congestive cardiomyopathy
  * left ventricular ejection fraction < 40% by multigated radionucleotide angiogram (MUGA), angiography, or echocardiography
  * coronary artery disease with continuing symptoms of angina pectoris
  * life-threatening cardiac arrhythmias
* Atrial septostomy within 1 year.
* History of pulmonary embolism prior to diagnosis of PAH unless it can be documented that chronic thromboembolic pulmonary hypertension (CTEPH) has been specifically excluded (e.g., ventilation/perfusion (VQ) scan, pulmonary angiogram).
* Restrictive lung disease: TLC < 60% of normal predicted value.
* Obstructive lung disease: forced expiratory volume/forced vital capacity (FEV1/FVC) < 0.5 or clinically relevant chronic obstructive lung disease or asthma (including any patient requiring concomitant medication to control symptoms of bronchospasm including as needed (p.r.n.) use).
* Clinically relevant bleeding disorder or active bleeding.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C or hepatic cirrhosis.
* Pregnant or breast-feeding.
* Chronic renal insufficiency, as defined by a creatinine of > 2.5 mg/dL or the requirement for dialysis.
* Hemoglobin < 75% of the lower limit of normal range.
* Any condition that prevents compliance with the protocol or adherence to therapy or ability to provide informed consent.
* Participation in any other clinical trial, except observational, or receipt of an investigational product within 30 days prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - University of South Alabama Medical, Mobile, Alabama
  - Arizona Pulmonary Associates, Ltd., Phoenix, Arizona
  - Kaiser Foundation Hospital, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Suncoast Lung Research, LLC, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Winthrop University Hospital, Mineola, New York
  - North Shore Long Island Jewish Health System, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracus, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - The Ohio State University, The Dorothy M. Davis Heart & Lung Research Institute, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center-Presbyterian, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - Central Utah Clinic, P.C., Provo, Utah
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Comprehensive Cardiovascular Care Group LLC, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 22 U.S. centers
Pre-assignment Details: Adults with pulmonary arterial hypertension (PAH) who were using Ventavis (Iloprost) Inhalation Solution Delivered by I-Neb Utilizing Power Disc-6 (PD-6) were enrolled
Groups:
- Iloprost: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-6 (PD-6) and Power Disc-15 (PD-15).
Period: Overall Study
Arm/Group | Iloprost
Started | 63
Completed | 34
Not Completed | 29
Not completed — Adverse Event | 12
Not completed — Investigator's judgement | 5
Not completed — Inhaled medication other than iloprost | 4
Not completed — Withdrawal of consent | 3
Not completed — Other | 3
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Iloprost
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Treatment-emergent Adverse Events (AEs)
Description: Number of patients reporting at least one treatment-emergent AE/Serious AE
Time Frame: From the first dose to last dose of investigational product, an average of approximately 268 days, plus 48 hours
Population: Safety population
Measure: Number; unit: participants
Groups:
- Iloprost: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-15 (PD-15).
Arm/Group | Iloprost
Number analyzed (Participants) | 63
participants | 53

2. Primary Outcome: Number of Patients Who Discontinued Iloprost PD-15 Treatment Due to an AE
Description: Number of patients reporting at least one treatment-emergent AE/Serious AE leading to discontinuation of study investigational treatment
Time Frame: From the first dose of investigational product to study discontinuation, an average of approximately 268 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 63
participants | 8

3. Primary Outcome: Number of Patients Reporting Treatment-emergent Serious AEs
Description: Number of patients reporting at least one treatment-emergent serious AEs
Time Frame: From the first to last dose of investigational product, an average of approximately 268 days, plus 48 hours
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 63
participants | 18

4. Primary Outcome: Systolic Blood Pressure - Iloprost PD-6 (Period 1)
Description: Systolic blood pressure was measured immediately prior to first dosing with Iloprost PD-15
Time Frame: Day 1
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Iloprost: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-6 (PD-6).
Arm/Group | Iloprost
Number analyzed (Participants) | 63
mmHg | 117.7 (15.61)

5. Primary Outcome: Systolic Blood Pressure - Iloprost PD-15 (Period 2)
Description: Systolic blood pressure was measured on Day 28 of treatment with Iloprost PD-15
Time Frame: Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 61
mmHg | 116.2 (14.71)

6. Primary Outcome: Systolic Blood Pressure - Iloprost PD-15 (Period 3)
Description: Systolic blood pressure was measured at the end of study visit
Time Frame: an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 53
mmHg | 119.0 (17.47)

7. Primary Outcome: Change in Systolic Blood Pressure - (Period 1 to Period 2)
Description: Systolic blood pressure was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and Day 28 of treatment with Iloprost PD-15 (Period 2)
Time Frame: Day 1 and Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 61
mmHg | -1.9 (13.07)

8. Primary Outcome: Change in Systolic Blood Pressure - (Period 1 to Period 3)
Description: Systolic blood pressure was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and at the end of treatment with Iloprost PD-15 (Period 3)
Time Frame: Day 1 and End of study visit, an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 53
mmHg | 0.8 (17.82)

9. Primary Outcome: Diastolic Blood Pressure - Iloprost PD-6 (Period 1)
Description: Diastolic blood pressure was measured immediately prior to first dosing with Iloprost PD-15
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 63
mmHg | 67.6 (10.57)

10. Primary Outcome: Diastolic Blood Pressure - Iloprost PD-15 (Period 2)
Description: Diastolic blood pressure was measured on Day 28 of treatment with Iloprost PD-15
Time Frame: Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 61
mmHg | 67.0 (8.86)

11. Primary Outcome: Diastolic Blood Pressure - Iloprost PD-15 (Period 3)
Description: Diastolic blood pressure was measured at the end of study visit
Time Frame: an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 53
mmHg | 65.6 (9.50)

12. Primary Outcome: Change in Diastolic Blood Pressure - (Period 1 to Period 2)
Description: Diastolic blood pressure was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and Day 28 of treatment with Iloprost PD-15 (Period 2)
Time Frame: Day 1 and Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 61
mmHg | -0.5 (9.66)

13. Primary Outcome: Change in Diastolic Blood Pressure - (Period 1 to Period 3)
Description: Diastolic blood pressure was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and at the end of treatment with Iloprost PD-15 (Period 3)
Time Frame: Day 1 and End of study visit, an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost
Number analyzed (Participants) | 53
mmHg | -2.3 (10.64)

14. Primary Outcome: Heart Rate - Iloprost PD-6 (Period 1)
Description: Heart rate was measured immediately prior to first dosing with Iloprost PD-15
Time Frame: Day 1
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost
Number analyzed (Participants) | 63
beats per minute | 73.8 (11.67)

15. Primary Outcome: Heart Rate - Iloprost PD-15 (Period 2)
Description: Heart rate was measured on Day 28 of treatment with Iloprost PD-15
Time Frame: Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost
Number analyzed (Participants) | 61
beats per minute | 74.2 (11.76)

16. Primary Outcome: Heart Rate - Iloprost PD-15 (Period 3)
Description: Heart rate was measured at the end of study visit
Time Frame: an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost
Number analyzed (Participants) | 53
beats per minute | 75.6 (13.66)

17. Primary Outcome: Change in Heart Rate - (Period 1 to Period 2)
Description: Heart rate was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and Day 28 of treatment with Iloprost PD-15 (Period 2)
Time Frame: Day 1 and Day 28
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost
Number analyzed (Participants) | 61
beats per minute | 0.3 (12.24)

18. Primary Outcome: Change in Heart Rate - (Period 1 to Period 3)
Description: Heart rate was measured on Day 1 prior to treatment with Iloprost PD-15 (Period 1) and at the end of treatment with Iloprost PD-15 (Period 3)
Time Frame: Day 1 and End of study visit, an average of approximately 268 days
Population: Safety population - missing data were not imputed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost
Number analyzed (Participants) | 53
beats per minute | 2.6 (13.89)

19. Secondary Outcome: Average Inhalation Time - Iloprost PD-6 (Period 1)
Description: The time and date of inhalation, inhalation time (minutes), and dose completion status (<12.5%, ≥12.5 to <100%, full) were recorded in the memory chip of the I-neb® AAD® each time it was used.
Time Frame: average of approximately 28 days
Population: Modified intent-to-treat (MITT) population - includes all enrolled patients without major protocol violations, who received at least one dose of iloprost with PD-15, and had one or more post-baseline evaluations for pharmacodynamic endpoints.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost
Number analyzed (Participants) | 58
minutes | 13.9 (5.83)

20. Secondary Outcome: Average Inhalation Time - Iloprost PD-15 (Period 2)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost
Number analyzed (Participants) | 58
minutes | 7.7 (4.01)

21. Secondary Outcome: Average Inhalation Time - Iloprost PD-15 (Period 3)
Description: as for outcome 19
Time Frame: average of approximately 240 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost
Number analyzed (Participants) | 49
minutes | 8.4 (4.30)

22. Secondary Outcome: Change in Average Inhalation Time - (Period 1 to Period 2)
Description: as for outcome 19
Time Frame: average approximately 56 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost
Number analyzed (Participants) | 58
minutes | -6.1 (2.92)
Statistical Analysis 1: Comparison: Iloprost; Comparison of the change in average inhalation times from Period I (PD-6) to Period II (PD-15); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -6.1, 95% CI 2-sided [-6.9 to -5.4]

23. Secondary Outcome: Average Number of Days of Dosing - Iloprost PD-6 (Period 1)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iloprost
Number analyzed (Participants) | 58
days | 27.6 (1.11)

24. Secondary Outcome: Average Number of Days of Dosing - Iloprost PD-15 (Period 2)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iloprost
Number analyzed (Participants) | 58
days | 27.4 (2.66)

25. Secondary Outcome: Average Number of Days of Dosing - Iloprost PD-15 (Period 3)
Description: as for outcome 19
Time Frame: average of approximately 240 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iloprost
Number analyzed (Participants) | 49
days | 240 (139.03)

26. Secondary Outcome: Change in Average Number of Days of Dosing - (Period 1 to Period 2)
Description: as for outcome 19
Time Frame: average approximately 56 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iloprost
Number analyzed (Participants) | 58
days | -0.2 (2.93)
Statistical Analysis 1: Comparison: Iloprost; Comparison of the change in average number of days of dosing from Period I (PD-6) to Period II (PD-15); Test type: Superiority or Other; p = 0.59, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.0 to 0.6]

27. Secondary Outcome: Average Number of Daily Doses - Iloprost PD-6 (Period 1)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | Iloprost
Number analyzed (Participants) | 58
doses per day | 5.1 (1.48)

28. Secondary Outcome: Average Number of Daily Doses - Iloprost PD-15 (Period 2)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | Iloprost
Number analyzed (Participants) | 58
doses per day | 5.6 (1.14)

29. Secondary Outcome: Average Number of Daily Doses - Iloprost PD-15 (Period 3)
Description: as for outcome 19
Time Frame: average of approximately 240 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | Iloprost
Number analyzed (Participants) | 49
doses per day | 4.7 (1.69)

30. Secondary Outcome: Change in Average Number of Daily Doses - (Period 1 to Period 2)
Description: as for outcome 19
Time Frame: average approximately 56 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | Iloprost
Number analyzed (Participants) | 58
doses per day | 0.5 (1.00)
Statistical Analysis 1: Comparison: Iloprost; Comparison of the change in average number of daily doses from Period I (PD-6) to Period II (PD-15); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [0.2 to 0.7]

31. Secondary Outcome: Percentage of Complete Doses Delivered - Iloprost PD-6 (Period 1)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost
Number analyzed (Participants) | 58
percentage of complete doses | 84.3 (23.42)

32. Secondary Outcome: Percentage of Complete Doses Delivered - Iloprost PD-15 (Period 2)
Description: as for outcome 19
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost
Number analyzed (Participants) | 58
percentage of complete doses | 95.4 (14.75)

33. Secondary Outcome: Percentage of Complete Doses Delivered - Iloprost PD-15 (Period 3)
Description: as for outcome 19
Time Frame: average of approximately 240 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost
Number analyzed (Participants) | 49
percentage of complete doses | 94.2 (12.02)

34. Secondary Outcome: Change in Percentage of Complete Doses Delivered - (Period 1 to Period 2)
Description: as for outcome 19
Time Frame: average approximately 56 days
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost
Number analyzed (Participants) | 58
percentage of complete doses | 11.0 (17.23)
Statistical Analysis 1: Comparison: Iloprost; Comparison of the change in percentage of complete doses delivered from Period I (PD-6) to Period II (PD-15); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 11.0, 95% CI 2-sided [6.5 to 15.6]

35. Secondary Outcome: New York Health Association (NYHA) Functional Class - Iloprost PD-6 (Period 1, Prior to First Dose With Iloprost PD-15)
Description: Disease severity was assessed by NYHA classification of PAH criteria: Class I: no limitation of physical activity (PA). Ordinary PA: no undue dyspnea/fatigue, chest pain, near syncope. Class II: slight limitation of PA. Comfortable at rest. Ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class III: marked limitation of PA. Comfortable at rest. Less than ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class IV: inability to carry out PA without symptoms. Right heart failure. Dyspnea/fatigue may even have been present at rest. Discomfort increased by any PA.
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 58
participants
  Class I | 3
  Class II | 17
  Class III | 34
  Class IV | 4

36. Secondary Outcome: NYHA Functional Class - Iloprost PD-15 (Period 2, Day 28)
Description: as for outcome 35
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 55
participants
  Class I | 3
  Class II | 17
  Class III | 33
  Class IV | 2

37. Secondary Outcome: NYHA Functional Class - Iloprost PD-15 (Period 3, End of Study Visit))
Description: as for outcome 35
Time Frame: average of approximately 268 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 48
participants
  Class I | 3
  Class II | 20
  Class III | 19
  Class IV | 6

38. Secondary Outcome: Number of Patients With Improved, no Change, or Worsening of NYHA Functional Class - (Period 1, Prior to First Dose With Iloprost PD-15 to Period 2, Day 28)
Description: as for outcome 35
Time Frame: average approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 55
participants
  Improved | 4
  No change | 50
  Worse | 1

39. Secondary Outcome: Number of Patients With Improved, no Change, or Worsening of NYHA Functional Class - (Period 1, Prior to First Dose With Iloprost PD-15 to Period 3, End of Study Visit)
Description: as for outcome 35
Time Frame: average approximately 268 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 48
participants
  Improved | 7
  No change | 37
  Worse | 4

40. Secondary Outcome: Patient Global Self Assessment - Iloprost PD-6 (Period 1, Prior to First Dose With Iloprost PD-15)
Description: The Patient Global Self Assessment is a 7-point scale that was presented to patients prior to conducting visit-specific study procedures. Patients were asked to compare their current PAH status to their status in the past by selecting one of the following options: markedly better; moderately better; mildly better; no change; mildly worse; moderately worse; or markedly worse.
  On Day 1 prior to their first dose of iloprost with PD-15 (Baseline), patients were asked to compare their PAH status to that during Screening (if the Screening and Baseline visits were conducted on the same day, then patients were asked to compare their PAH status to that in the past 2 weeks). On Day 28 and at the end of study (EOS) visit, patients were asked to compare their PAH status to that of the previous visit.
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 58
participants
  Markedly better | 8
  Moderately better | 8
  Mildly better | 9
  No change | 31
  Mildly worse | 2
  Moderately worse | 0
  Markedly worse | 0

41. Secondary Outcome: Patient Global Self Assessment - Iloprost PD-15 (Period 2, Day 28)
Description: The Patient Global Self Assessment is a 7-point scale that was presented to patients prior to conducting visit-specific study procedures. Patients were asked to compare their current PAH status to their status in the past by selecting one of the following options: markedly better; moderately better; mildly better; no change; mildly worse; moderately worse; or markedly worse.
  On Day 1 prior to their first dose of iloprost with PD-15 (Baseline), patients were asked to compare their PAH status to that during Screening (if the Screening and Baseline visits were conducted on the same day, then patients were asked to compare their PAH status to that in the past 2 weeks). On Day 28 and at the EOS visit, patients were asked to compare their PAH status to that of the previous visit.
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 56
participants
  Markedly better | 7
  Moderately better | 15
  Mildly better | 12
  No change | 21
  Mildly worse | 0
  Moderately worse | 1
  Markedly worse | 0

42. Secondary Outcome: Patient Global Self Assessment - Iloprost PD-15 (Period 3, End of Study Visit))
Description: as for outcome 41
Time Frame: average of approximately 268 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 50
participants
  Markedly better | 6
  Moderately better | 10
  Mildly better | 11
  No change | 17
  Mildly worse | 4
  Moderately worse | 1
  Markedly worse | 1

43. Secondary Outcome: Number of Patients With Improved, no Change, or Worse Patient Global Self Assessment - Change From Previous Visit to Period 2, Day 28
Description: as for outcome 41
Time Frame: average of approximately 28 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 56
participants
  Improved | 34
  No change | 21
  Worse | 1

44. Secondary Outcome: Number of Patients With Improved, no Change, or Worse Patient Global Self Assessment - Change From Previous Visit to Period 3, End of Study Visit
Description: as for outcome 41
Time Frame: average of approximately 268 days
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 50
participants
  Improved | 27
  No change | 17
  Worse | 6

ADVERSE EVENTS:
Time Frame: From the first to last dose of investigational product, an average of approximately 268 days, plus 48 hours
Description: Serious treatment-emergent adverse events
Arm/Group | Iloprost
Serious Adverse Events (participants affected / at risk) | 18/63
Other Adverse Events (participants affected / at risk) | 50/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost (N=63)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Carotid artery disease (Nervous system disorders) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Chest pain (General disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mental status changes (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost (N=63)
ANAEMIA (Blood and lymphatic system disorders) | 4
PALPITATIONS (Cardiac disorders) | 5
VERTIGO (Ear and labyrinth disorders) | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 9
NAUSEA (Gastrointestinal disorders) | 9
CHEST PAIN (General disorders) | 4
FATIGUE (General disorders) | 10
OEDEMA (General disorders) | 4
ACUTE SINUSITIS (Infections and infestations) | 3
BRONCHITIS (Infections and infestations) | 5
SINUSITIS (Infections and infestations) | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9
URINARY TRACT INFECTION (Infections and infestations) | 6
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3
GOUT (Metabolism and nutrition disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 4
DIZZINESS (Nervous system disorders) | 8
HEADACHE (Nervous system disorders) | 11
ANXIETY (Psychiatric disorders) | 4
INSOMNIA (Psychiatric disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3
HAEMATOMA (Vascular disorders) | 4
HYPERTENSION (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No